CLINICAL TRIAL: NCT05648604
Title: An Adapted Evidenced-Based Mentored Community Gardening Intervention for Skin Cancer Survivors: A Single-Arm Feasibility Study (Harvest for Health Together Arizona)
Brief Title: Mentored Community Gardening for Individuals With Skin Cancer
Acronym: H4H2-AZ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: Banner University Medical Center (Other)
Responsible Party: Principal Investigator, Meghan Skiba, Assistant Professor, University of Arizona
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 00002169
Record Dates: First submitted 2022-11-18; First posted 2022-12-13 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Melanoma; Cancer Survivorship; Skin Cancer; Basal Cell Carcinoma; Squamous Cell Carcinoma; Melanoma (Skin)
Keywords: Nutrition; UV; Physical Activity; Gardening
MeSH Terms: conditions — Melanoma; Skin Neoplasms; Carcinoma, Basal Cell; Carcinoma, Squamous Cell; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Mentored Community Gardening (Experimental): This arm will consist of gardening at least once per week, meeting with a master gardener mentor bi-monthly, and attending a gardening informational workshop once monthly.
  Interventions: Behavioral: Mentored Community Gardening

INTERVENTIONS:
Behavioral: Mentored Community Gardening — This arm will consist of gardening at least once per week, meeting with a master gardening mentor twice monthly, and attending a gardening informational workshop once monthly.

SUMMARY:
The investigators will conduct a single-arm pilot feasibility trial of mentored community gardening for melanoma survivors integrating dosimeters and accelerometers. Harvest for Health Together Arizona (H4H2-AZ) is an evidence-based program adapted for arid desert gardening that also addresses sun safety through group workshops and peer education. The primary aim is to evaluate adherence to the intervention.

DETAILED DESCRIPTION:
In collaboration with Banner Health, University of Arizona Cancer Center, Community Gardens of Tucson, and UArizona Pima County Cooperative Extension Master Gardeners, the investigators will conduct a pilot feasibility study of community gardening in melanoma survivors integrating UV sensors. Harvest for Health Together Arizona (H4H2-AZ) is an evidence-based program adapted for arid desert gardening that also addresses sun safety through experiential workshops and education. The investigators propose to evaluate adherence to and acceptability of the intervention. The investigators aim to see if H4H2-AZ may improve cancer preventive health behaviors (including diet, physical activity, energy balance, and UV protection) and quality of life among melanoma survivors.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older at their last birthday & in good general health.
* Clinical diagnosis of skin cancer (including in situ).
* Has access to a phone or tablet with a camera and internet.
* Currently living in Pima County Arizona.
* Ability to understand and speak English.
* Ability to provide written informed consent document.
* Ability to physically participate in gardening activities (including kneeling, sitting, bending, and carrying up to 10 pounds) with or without the use of mobility assistive devices.

Exclusion Criteria:

* Currently immunosuppressed by virtue of medication or disease.
* Has a diagnosed and uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2023-02-02 (Actual); Primary Completion 2024-12-15 (Actual); Study Completion 2024-12-15 (Actual)

PRIMARY OUTCOMES:
Mean number of scheduled sessions a participant attends during intervention | 6 months
  Adherence will be measured by attendance to the number of sessions (including weekly gardening, meetings with mentors, and group workshops) a participant attends.

SECONDARY OUTCOMES:
UV Exposure | 6 months
  Dosimeter (Scienterra) measured cumulative UV exposure [Units: Watts per square meter (W/m^2), UV Index (UVI), Standard Erythema Dose (SED), or Minimal Erythema Dose (MED)]
Fruit and Vegetable Servings | 6 months
  Dietary fruit and vegetable intake (average total servings/day) assessed by 24-hour dietary recall
Total sedentary time | 6 months
  Sedentary time (inactive minutes/day) measured by accelerometer (Actigraph Link GT9X)

OTHER OUTCOMES:
Health Related Quality of Life (HR-QOL) | 6 months
  Functional Assessment of Cancer Therapy - Melanoma (FACT-M) is a melanoma specific questionnaire which will measure HR-QOL in participants. Items are measured on a 0-4 Likert scale.The FACT-M consists of 51 items with a total score ranging from 0-204. A higher score indicates better HR-QOL.
Average acceptability of intervention | 6 months
  Acceptability of intervention and sensors will be assessed using the Acceptability of Intervention Measure which includes 12 items on a 1-5 scale and summed. Scores range 12-60; higher scores reflect greater acceptability.

CONTACTS AND LOCATIONS:
Overall Officials: Meghan B Skiba, PhD, Principal Investigator — University of Arizona College of Nursing
Locations (1):
- University of Arizona Cancer Center, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Skiba MB, Miller D, Stratton DB, Hall CA, McKenna S, Blair CK, Demark-Wahnefried W. Adaptation and study protocol for harvest for health together Arizona: A mentored community garden intervention for survivors of cancer. Contemp Clin Trials Commun. 2024 Mar 28;39:101290. doi: 10.1016/j.conctc.2024.101290. eCollection 2024 Jun. PMID 38595771